CLINICAL TRIAL: NCT07291219
Title: Registry of Pavia Chronic Heart Failure Patients-observational Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Stefano Ghio, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: CHF_22
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years

SUMMARY:
Registry of Pavia chronic heart failure patients-observational study

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent to participate for the prospective evaluations
* Suffer from CHF
* Be aged 18 years and over

Exclusion Criteria:

* Withdrawn of the consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All ambulatory patients with HF in follow up at Fondazione IRCCS Policlinico San Matteo will be prospectively included in this study.
Sampling Method: Probability Sample
Enrollment: 101 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
accurate and comprehensive data collection for all types of diseases that manifest themselves with heart failure in order to verify the "trajectory" of the disease | From enrollment to the end of treatment at visit 11 (9th years)
  More specifically, mortality will be assessed one, five, and ten years after the initial diagnosis of heart failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Pavia, Italy